CLINICAL TRIAL: NCT03798275
Title: The Effect of Coffee Consumption on Fetal Renal Artery Blood Flow and Amniotic Fluid Volume in the Third Trimester of Pregnancy
Brief Title: Coffee Consumption and Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf MADENDAG, obstetrics and gynecology, Kayseri Education and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/489
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Coffee; Pregnancy
Keywords: amniotic fluid index; caffeine; coffee; oligohydramnios
MeSH Terms: conditions — Oligohydramnios | interventions — Coffee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the study group (Active Comparator): healthy pregnant women with borderline oligohydramnios who accept to drink a cup of coffee
  Interventions: Dietary Supplement: coffee
- the control group (No Intervention): healthy pregnant women with normal amniotic volume

INTERVENTIONS:
Dietary Supplement: coffee — 2 g Nescafe Clasico contains approximately 65 mg caffeine
  Arms: the study group

SUMMARY:
Coffee, tea, and cocoa contain caffeine, a plant alkaloid. They are frequently consumed during pregnancy. We examined the effect of coffee consumption on fetal renal artery blood flow and amniotic fluid index (AFI) in the third trimester of pregnancy

DETAILED DESCRIPTION:
This cross-sectional study occurred in a tertiary center with volunteer pregnant women who agreed to drink coffee. In healthy pregnant women with isolated borderline oligohydramnios, AFI and fetal renal artery blood flow indices were evaluated before and after coffee consumption. Sixty three patients for the borderline oligohydramnios group (the study group) were included in this study. These patients were compared with 63 healthy pregnant women who had normal amniotic fluid volume (the control group)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a singleton, uncomplicated pregnancy between the 34th and 37th weeks of gestation were included in this study during routine antenatal examinations

Exclusion Criteria:

* abnormal amniotic fluid volume (AFV), any intake of nutrient or fluid within the 4 hours previous to ultrasonographic examination [10], abnormal Doppler blood flow, hypertension, preeclampsia, chromosomal anomaly, intrauterine growth restriction, fetal anomaly, collagen vascular disease, ruptured fetal membranes, and multiple pregnancies.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
amniotic fluid index | two hours
fetal renal artery doppler indices | two hours

CONTACTS AND LOCATIONS:
Overall Officials: YUSUF MADENDAĞ, Principal Investigator — Sağlık Bilimleri Üniversitesi Kayseri Şehir hastanesi
Locations (1):
- Yusuf Madendağ, Kayseri, Turkey (Türkiye)